CLINICAL TRIAL: NCT00028561
Title: A Phase I Study of Epothilone B Analog BMS 247550 in Combination With Carboplatin in Recurrent and/or Refractory Solid Tumors
Brief Title: BMS-247550 Plus Carboplatin in Treating Patients With Recurrent or Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02726; 12657; CDR0000069105 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — ixabepilone; Carboplatin

ARMS (1):
- Treatment (ixabepilone, carboplatin) (Experimental): Patients receive BMS-247550 IV over 1 hour on days 1, 8, and 15 followed by carboplatin IV over 1 hour on day 1. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with a CR receive 2 additional courses after achieving CR or up to a total of 6 courses
  Interventions: Drug: ixabepilone; Drug: carboplatin; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of BMS-247550 when given together with carboplatin in treating patients with recurrent or refractory solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of BMS-247550 when given in combination with carboplatin in patients with recurrent or refractory solid tumors.

II. Determine the dose-limiting toxicity and safety of this regimen in these patients.

III. Determine the plasma pharmacokinetics of this regimen in these patients. IV. Determine, preliminarily, any antitumor activity of this regimen in these patients.

V. Correlate the protein expression of survivin with the expression of other apoptotic regulators, the apoptotic index, and response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of BMS-247550.

Patients receive BMS-247550 IV over 1 hour on days 1, 8, and 15 followed by carboplatin IV over 1 hour on day 1. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 2 additional courses after achieving CR or up to a total of 6 courses. The first two cohorts of 3-6 patients each receive escalating doses of BMS-247550 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT).The third and fourth cohorts of 10 patients each receive escalating doses of BMS-247550 until the MTD is determined. The MTD is defined as the dose preceding that at which at least 3 of 10 patients experience DLT. Once the MTD is determined for the third and fourth cohorts, 15 additional patients are treated at the MTD. Patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective
* Measurable or evaluable disease
* Lesion accessible for core or excisional biopsy if being treated at the maximum tolerated dose (MTD)

  * No biliary tract dilation if radiologically guided biopsy of the liver is planned
  * No requirement for core biopsy of lung lesion that is not pleural based
  * No requirement for laparotomy or thoracotomy solely for biopsy
  * No medical condition that would preclude biopsy
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - ECOG 0-1 if being treated at the MTD
* More than 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No prior bleeding disorder or unexplained bleeding if being treated at the MTD
* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* PT/PTT normal
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent uncontrolled illness that would preclude study participation
* No ongoing or active infection
* No grade 2 or greater neuropathy (sensory or motor)
* No prior severe allergic reaction attributable to compounds containing Cremophor EL or platinum agents
* No psychiatric illness or social situation that would preclude study compliance
* No medical condition that would preclude study if being treated at the MTD
* At least 4 week since prior immunotherapy
* At least 24 hours since prior growth factors
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No more than 3 prior chemotherapy regimens
* No prior epothilone agents
* At least 1 week since prior hormonal therapy directed at malignancy
* Concurrent hormone replacement therapy allowed
* At least 4 weeks since prior wide-field radiotherapy involving 30% or more of bone marrow
* See Disease Characteristics
* At least 4 weeks since prior investigational agents
* No prior or concurrent St. John's Wort
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent heparin or other anticoagulants if being treated at the MTD
* No concurrent inhibitors of cytochrome P450 3AP (CYP3A4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2001-10; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
MTD of ixabepilone defined as the first dosage tier below the MAD in which =< 1/6 patients experiences a DLT | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics of ixabepilone and carboplatin | Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sullivan, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States